CLINICAL TRIAL: NCT04683185
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple Ascending Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of E6742 in Japanese Healthy Adult Subjects
Brief Title: A Study to Assess the Safety and Tolerability of E6742 in Japanese Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: E6742-J081-005; jRCT2031200316 (Registry Identifier: jRCT)
Record Dates: First submitted 2020-12-21; First posted 2020-12-24 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-05

CONDITIONS: Healthy Volunteers
Keywords: E6742; Healthy participants; Pharmacokinetics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 2: E6742 200 mg or Placebo (Experimental): Participants will receive E6742 200 mg or E6742-matched placebo, tablets, orally, twice daily for 6 days under fasted conditions and once on Day 7 in the morning.
  Interventions: Drug: E6742; Drug: Placebo
- Cohort 3: E6742 400 mg or Placebo (Experimental): Participants will receive E6742 400 mg or E6742-matched placebo, tablets, orally, twice daily for 6 days under fasted conditions and once on Day 7 in the morning.
  Interventions: Drug: E6742; Drug: Placebo
- Cohort 1: E6742 100 milligram (mg) or Placebo (Experimental): Participants will receive E6742 100 mg or E6742-matched placebo, tablets, orally, twice daily for 6 days under fasted conditions and once on Day 7 in the morning.
  Interventions: Drug: E6742; Drug: Placebo

INTERVENTIONS:
Drug: E6742 — E6742 tablets.
Drug: Placebo — E6742-matched placebo tablets.

SUMMARY:
The primary purpose of the study is to evaluate the safety, tolerability and pharmacokinetics (PK) of multiple ascending oral doses of E6742 in Japanese healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

1. Non-smoking, male or female Japanese, greater than or equal to (>=) age 20 years and less than or equal to (<=) 55 years old at the time of informed consent
2. Body mass index (BMI) >=18.5 and less than (<) 25.0 kilogram per meter square (kg/m^2) at Screening

Exclusion Criteria:

1. Females who are breastfeeding or pregnant at Screening or Baseline
2. Females of childbearing potential who:

   * Within 28 days before study entry, did not use a highly effective method of contraception, which includes any of the following:

     * Total abstinence
     * An intrauterine device (IUD) or intrauterine hormone-releasing system (IUS)
     * A contraceptive implant
     * An oral contraceptive
     * Have a vasectomized partner with confirmed azoospermia
   * Do not agree to use a highly effective method of contraception (as described above) throughout the entire study period and for 28 days after study drug discontinuation
3. Males who have not had a successful vasectomy (confirmed azoospermia) or they and their female partners do not meet the criteria above (that is, not of childbearing potential or practicing highly effective contraception throughout the study period and for 5 times the half-life of the study drug plus 90 days after study drug discontinuation)
4. Clinically significant illness that requires medical treatment within 8 weeks or a clinically significant infection within 4 weeks before dosing
5. Any history of gastrointestinal surgery that may affect PK profiles of E6742 at Screening
6. Any clinically abnormal symptom or organ impairment found by medical history, ophthalmic examination or chest X ray test at Screening, or founded by physical examinations, vital signs, ECG finding, or laboratory test results at Screening or Baseline
7. A prolonged QTc corrected using Fridericia's method (QTcF) interval (QTcF greater than [>] 450 millisecond [ms]) demonstrated on ECG at Screening or Baseline. A history of risk factors for torsade de pointes or the use of concomitant medications that prolonged the QT/QTc interval
8. Persistent systolic blood pressure >130 millimeter of mercury (mmHg) or diastolic blood pressure >85 mmHg diastolic at Screening or Baseline
9. Heart rate less than 45 or more than 100 beats per min at Screening or Baseline
10. Any lifetime history of suicidal ideation or any lifetime history of suicidal behavior as indicated by the Suicidal Ideation section of the Columbia Suicide Severity Rating Scale (C-SSRS)
11. Any lifetime history of psychiatric disease
12. Any current psychiatric symptoms as indicated by a standard screening tool (Patient Health Questionnaire 9 [PHQ 9])
13. Any suicidal ideation with intent with or without a plan within Screening or 6 months before Screening (that is, answering "Yes" to questions 4 or 5 on the C-SSRS)
14. History of autoimmune disease or immunodeficiency
15. Known to be positive for tuberculosis test (T-spot. TB Test) at Screening
16. Received immunoglobulin or blood preparation within 6 months before the study treatment
17. Received inoculation within 4 weeks before the study treatment (8 weeks before in case of live or attenuated vaccine)
18. Family living together or cohabitant of a patient with an influenza virus infection
19. In contact with Coronavirus disease (COVID 19) patient within 4 weeks before study drug administration
20. Known to be other than negative for Severe acute respiratory syndrome coronavirus 2 (SARS Cov 2) antibody test at Screening
21. Known to be other than negative for SARS Cov 2 polymerase chain reaction (PCR) test at Screening or Baseline
22. History of retinopathy, maculopathy or macular degeneration

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-12-28 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2021-06-21 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Baseline up to 28 days after the last dose of study drug (approximately Day 35)
  Safety assessments will consist of monitoring and recording all adverse events (AEs) and SAEs; laboratory evaluation for hematology, blood chemistry, and urine values; periodic measurement of vital signs and electrocardiograms (ECGs); and the performance of physical examinations.
Cmax: Maximum Observed Plasma Concentration for E6742 and its Metabolite (ER-001132963) on Day 1 | Day 1: 0-12 hours
tmax: Time at Which the Highest Drug Plasma Concentration Occurs for E6742 and its Metabolite (ER-001132963) on Day 1 | Day 1: 0-12 hours
AUC(0-12h): Area Under the Plasma Concentration-time Curve From Zero Time to 12 Hours Postdose for E6742 and its Metabolite (ER-001132963) on Day 1 | Day 1: 0-12 hours
AUC Metabolite to E6742 Ratio Following Molecular Weight Correction to E6742 Equivalents on Day 1 | Day 1: 0-12 hours
Css,max: Maximum Observed Plasma Concentration at Steady State for E6742 and its Metabolite (ER-001132963) on Day 7 | Day 7: 0-168 hours
tss,max: Time at Which the Highest Drug Plasma Concentration Occurs at Steady State for E6742 and its Metabolite (ER-001132963) on Day 7 | Day 7: 0-168 hours
Css,av: Average Steady State Plasma Concentration for E6742 and its Metabolite (ER-001132963) on Day 7 | Day 7: 0-168 hours
AUC(0-t): Area Under the Plasma Concentration-time Curve From Zero Time to Time of Last Quantifiable Concentration for E6742 and its Metabolite (ER-001132963) on Day 7 | Day 7: 0-168 hours
AUC(0-12hr): Area Under the Plasma Concentration-time Curve Within a Dosing Interval at Steady State for E6742 and its Metabolite (ER-001132963) on Day 7 | Day 7: 0-12 hours
t1/2: Terminal Elimination Phase Half-life for E6742 and its Metabolite (ER-001132963) on Day 7 | Day 7: 0-168 hours
CLss/F: Apparent Total Clearance at Steady State for E6742 on Day 7 | Day 7: 0-168 hours
Vss/F: Apparent Volume of Distribution at Steady State for E6742 on Day 7 | Day 7: 0-168 hours
PTF: Peak-trough Fluctuation for E6742 and its Metabolite (ER-001132963) on Day 7 | Day 7: 0-168 hours
Accumulation Ratio for Cmax and AUC for E6742 and its Metabolite (ER-001132963) on Day 7 | Day 7: 0-168 hours
Metabolite to E6742 AUC Ratio Following Molecular Weight Correction to E6742 Equivalents on Day 7 | Day 7: 0-168 hours
AUC(0-12hr)ss: Area Under the Plasma Concentration-time Curve Within a Dosing Interval at Steady State for E6742 and its Metabolite (ER-001132963) on Day 7 | Day 7: 0-12 hours

SECONDARY OUTCOMES:
Change From Baseline in Corrected QT Interval (QTc) for E6742 | Day 1 and 7: 0-12 hours
  High precision method QT analysis (HPQT) will be performed using data extracted from the 12-hour holter recording obtained from the morning of day 1 (predose) through 12 hours after dosing, the morning of day 7 (predose) through 12 hours after dosing.

CONTACTS AND LOCATIONS:
Locations (1):
- Eisai Trial Site #1, Bunkyō-Ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.

REFERENCES:
- See also: Study results will be disclosed on the jRCT registry record. — https://jrct.niph.go.jp/en-latest-detail/jRCT2031200316